CLINICAL TRIAL: NCT00149305
Title: Genetic Study of Nephrolithiasis in Gouty Diathesis
Status: Terminated | Type: Observational
Why Stopped: Non significative preliminary data
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: GOUTY DIATESIS
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2009-10

CONDITIONS: Nephrolithiasis
Keywords: Gouty diathesis; Acid uric nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Genetic Linkage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood on EDTA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with gouthy diathesis
  Interventions: Other: Genetic analyses
- Healthy subjects
  Interventions: Other: Genetic analyses

INTERVENTIONS:
Other: Genetic analyses
  Groups: Patients with gouthy diathesis
Other: Genetic analyses
  Groups: Healthy subjects

SUMMARY:
Gouty diathesis describes uric acid or calcium oxalate nephrolithiasis and low urinary pH (<5.5). A hereditary component has been outlined for several forms of nephrolithiasis (such as hypercalciuria, hyperoxaluria, cystinuria, renal tubular acidosis), leading to the hypothesis of a genetic predisposition to nephrolithiasis. At the Unit of Nephrology, Ospedali Riuniti di Bergamo, more than 100 patients affected by gouty diathesis are followed. Fifty percent of them has a familiarity for kidney stones formation. The aim of our study is to identify the genetic factors that predispose to the development of nephrolithiasis in patients with gouty diathesis.

DETAILED DESCRIPTION:
INTRODUCTION Nephrolithiasis is a common disorder with a reported incidence of 12% in industrialized countries. The peak incidence is in ages 20s to 40s. Men are affected two to three times more often than women. Gouty diathesis describes uric acid or calcium oxalate nephrolithiasis and low urinary pH (<5.5) in the absence of excessive gastrointestinal alkali loses or dietary animal protein excess. Hyperuricemia, hypertriglyceridemia, and a history of gouty arthritis may be present. Subjects with gout are singularly predisposed to stone formation. Persistent acidity of the urine is a common manifestation of primary gout, that may be accompanied by uric acid nephrolithiasis. In the presence of an increase in the concentration of uric acid in the urine, the formation of uric acid stones is further facilitated.

In the primary forms of nephrolithiasis the most important predisposing factors for kidney stones are: hypercalciuria, hyperoxaluria, hyperuricosuria, hypocitraturia, hypomagnesuria, high urinary sulfate, low urine volume, high urinary sodium, cystinuria, infection, persistently high or low urinary pH. A hereditary component has been outlined for several of these abnormalities, leading to the hypothesis of a genetic predisposition to nephrolithiasis. Pirastu and co-workers took advantage from a small, isolated population from Sardinia, characterized by a high prevalence of Uric Acid Nephrolithiasis (UAN). The disease shows familial clustering, although the transmission of UAN does not follow a simple mendelian inheritance pattern, suggesting that hereditary factors could play an important role in susceptibility to UAN. They found an association of UAN to a new gene, called ZNF365, and in particular to its variant Ala62Thr, making it a strong candidate predisposing factor.

At the Unit of Nephrology, Ospedali Riuniti di Bergamo, we follow at the moment 560 patients with nephrolithiasis of which more than 100 are affected by gouty diathesis. 50% of all patients with gouty diathesis has a familiarity for kidney stones formation.

Understanding of the genetic factors that contribute to the development of this disorder may lead to earlier diagnosis, thus allowing to identify, within a family, subjects that are at risk to develop nephrolithiasis before manifestation of the disease. These subjects may have access to counseling aimed at modifying their dietetic and sanitary attitudes and/or to pharmacological treatments in order to prevent the manifestation of the renal disease or to slow its progression.

AIM The study is aimed at identifying the genetic factors that predispose to the development of nephrolithiasis in patients with gouty diathesis.

DESIGN Fifteen consecutive unrelated patients with familial form of nephrolithiasis associated with gouty diathesis (at least two affected subjects within a family) will be recruited, within 3 years, through the stone clinic ambulatory of the Unit of Nephrology, Ospedali Riuniti di Bergamo.

All patients affected by gouty diathesis and their selected relatives will undergo to the following evaluations:

* clinical history collection;
* renal ultrasound examination, to confirm previous diagnoses and identify asymptomatic cases;
* metabolic analyses, including:
* blood collection in order to evaluate: urate, urea triglycerides, calcium, phosphate, creatinine, bicarbonate, sodium, potassium, chloride, glucose;
* 24 hours urine collection in order to evaluate urate, calcium, phosphate, oxalate, citrate, urea, magnesium, sodium, chloride, creatinine, sulphate, ammonium; determination of urinary pH and titrable acidity; calculation of acid net excretion;
* morning urine spot in order to evaluate volume, pH, calcium, uric acid, creatinine;
* genetic analyses: 10 ml blood on EDTA to obtain DNA and 3 ml without anticoagulant to obtain serum from each subject will be collected.

ELIGIBILITY:
Inclusion Criteria:

* male and female, ≥ 10 years of age
* uric acid or calcium oxalate nephrolithiasis
* urinary 24 h pH < 5.5 in absence of high animal protein intake (urinary sulphate excretion <25 mM/24 h after one week of low animal protein intake)
* familial history of kidney stones (at least two first or second degree family members affected)
* written informed consent according to the Declaration of Helsinki guidelines

Exclusion Criteria:

* renal colic in the 4 weeks preceding evaluations
* excessive gastrointestinal alkali loses
* inability to fully understand the purposes of the study or to provide a written informed consent

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Unrelated patients with familial form of nephrolithiasis associated with gouty diathesis (at least two affected subjects within a family).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Daina, MD, Principal Investigator — Mario Negri Institute
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy